CLINICAL TRIAL: NCT01139034
Title: Rehabilitation Robot for Upper Limbs, Component Project 2: Hybrid of FES and Rehabilitation Robot for Treatment of Shoulder Subluxation
Brief Title: A Pilot Study of Shoulder Subluxation Treatment by Using the Self-Designed Surface Functional Electrical Stimulator
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Jin-Shin Lai, Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201002029D
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- shoulder FES treatment (Experimental)
  Interventions: Device: Self-designed surface functional electrical stimulator

INTERVENTIONS:
Device: Self-designed surface functional electrical stimulator — Use the self-designed surface functional electrical stimulator to improve the shoulder joint subluxation.
  Other Names: Self-designed surface functional electrical stimulation

SUMMARY:
The purpose of this study is to investigate the effects of the self-designed surface functional electrical stimulator on shoulder joint subluxation for stroke patients

DETAILED DESCRIPTION:
Functional electrical stimulation (FES) is a common and effective therapeutic approach for clinical treatments of shoulder subluxation. By applying low-frequency electrical stimulation to the target muscle groups, improvements may be observed in terms of muscle strength, subluxation, and passive humeral lateral rotation of the shoulder joint. In order to overcome issues regarding the integration of an FES and a rehabilitation robot, group members have designed a customized FES system approved by medical safety regulations. Despite sharing identical specifications with commercial models, the approved 2-channel FES system provides better integrity and control when working with the upper extremity rehabilitation robot. In this study, three patients with unilateral shoulder subluxation will be recruited. Limited shoulder x-ray photos shall be taken before, during, and after the FES shoulder subluxation treatment for studying the effects.

ELIGIBILITY:
Inclusion Criteria:

* stroke (1-3 months)
* Brunnstrom Stage I-III
* single, unilateral

Exclusion Criteria:

* aphasic
* shoulder impairment
* severe osteoporosis
* cardiac arrhythmias or having a pacemaker implanted
* abnormal cutaneous sensation at the target areas

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-12 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Upward migration index | 1 year

SECONDARY OUTCOMES:
Acromiohumeral distance | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shin Lai, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, NTUH, Taipei, Taiwan
Locations (1):
- Department of Physical Medicine and Rehabilitation, NTUH, Taipei, Taiwan